CLINICAL TRIAL: NCT01428505
Title: A Study to Characterize the Novel TSPO PET Radioligand [18F]PBR111 as an in Vivo Marker of Microglial Activation in Multiple Sclerosis
Brief Title: [18F]PBR111 and Microglial Activation in Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Study was terminated because there was insufficient data to complete the study objectives
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 115241
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 2-(6-chloro-2-(4-(3-fluoropropoxy)phenyl)imidazo(1,2-a)pyridin-3-yl)-N,N-diethylacetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no treatment (Other)
  Interventions: Radiation: [18F]PBR111

INTERVENTIONS:
Radiation: [18F]PBR111 — radioligand to assess binding to TSPO

SUMMARY:
This is a study aimed to characterize [18F]PBR111 as an in vivo marker of microglial activation in Multiple Sclerosis. Regional binding of [18F]PBR111 will be quantified with PET in the brain of up to 24 patients with multiple sclerosis and up to 24 age- and gender- matched healthy volunteers.

DETAILED DESCRIPTION:
Multiple Sclerosis is characterized by brain areas of focal neuroinflammation. Imaging of microglia activation in multiple sclerosis could represent a useful marker of neuroinflammation. A novel PET tracer with high affinity to TSPO, [18F]PBR111, is a promising tool for PET imaging of activated microglia.

This is a study aimed to characterize [18F]PBR111 as an in vivo marker of microglial activation in Multiple Sclerosis. Regional binding of [18F]PBR111 will be quantified with PET in the brain of up to 24 patients with multiple sclerosis and up to 24 age- and gender- matched healthy volunteers. A subgroup of patients and healthy volunteers will be scanned twice in consecutive days, to test the reproducibility of the measure. Another subgroup of patients will be re-scanned with [18F]PBR111 after 4-6 months. MRI-based measures will be acquired at baseline and, in those patients with later repeat PET scans, also after 4-6 months.

Data from this study will inform about the possible implementation of the [18F]PBR111 ligand to monitor the neuroinflammatory process, disease progression, and response to treatment in MS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged 20-70
2. Able to read, comprehend and record information written in English.
3. Capable of giving written informed consent
4. Provide a venous blood sample that will be used for genetics research and the in vitro ligand binding assay.
5. A female subject is eligible to participate if she is willing to follow contraception guidelines or if she is of non-childbearing potential.
6. Male subjects must agree to use one of the contraception methods

MS subjects:

1. Clinical or clinical and laboratory supported diagnosis of multiple sclerosis
2. EDSS score up to and including 7.5 at screening evaluation

Healthy Volunteers:

1. Healthy control subjects defined as free from clinically significant active disease as assessed by the Principal Investigator from their medical and psychiatric past and present history

-

Exclusion Criteria:

1. If female, positive urine pregnancy test
2. An estimated glomerular filtration rate (eGFR) of less than 60 ml/kg/1.73m2
3. History or presence of a neurological diagnosis
4. Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with radiation exposure.
5. Family history of cancer (one or more first-degree relative diagnosed before the age of 55).
6. Subject or caregiver is an immediate family member or employee of the participating Investigator, any of the participating site staff or GSK staff.
7. Any subject the investigator deems unsuitable for the study (e.g., due to either medical reasons, laboratory abnormalities or subject's unwillingness to comply with all study-related procedures).
8. Contraindications to MRI scanning
9. Any physical abnormality or functional disability which prevents the subject from acquiring a suitable position for scanning.
10. History of or suffers from claustrophobia or feels that he will be unable to lie still on his back in the PET camera or MRI scanner for a period of at least 90mins.
11. Unwillingness or inability to follow the procedures outlined in the protocol. -

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
VT of [18F]PBR111 | day 30
  Regional VT of [18F]PBR111 at baseline in MS patients and age- , gender-, and TSPO binding profile- matched healthy controls

SECONDARY OUTCOMES:
Test-retest variability of regional [18F]PBR111 | 8 months
  Test-retest variability of regional [18F]PBR111 VT in 2 consecutive days in MS patients and age- ,gender-, and TSPO binding profile- matched healthy controls
regional [18F]PBR111 VT | 1.5 years
  Change in regional [18F]PBR111 VT over ~ 4 months after a baseline assessment in MS patients
White matter lesion load and distribution | 1.5 years
  White matter lesion load (volume of pathological tissue) and distribution as measured by Gadolinium-enhanced and T2-weighted MRI in MS patients
Cortical grey matter lesion load and distribution | 1.5 years
  Cortical grey matter lesion load and distribution as estimated by the appropriate MRI technique (including high-field MRI in some cases)
Genetic polymorphisms related to the TSPO gene | 1.5 years
  Genetic polymorphisms related to the TSPO gene and/or genes encoding other proteins which may modulate the binding of ligands to TSPO or TSPO function

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, London, United Kingdom